CLINICAL TRIAL: NCT06850480
Title: A Multicenter, Randomized, Double-blind, Double-simulated, Positive Parallel-control Phase III Clinical Trails of JP-1366（Zastaprazan Citrate） Tablets and Nexium® on Reflux Esophagitis
Brief Title: A Phase III Clinical Trial for Efficacy and Safety Evaluation of JP-1366 Tablets on Reflux Esophagitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LZ031-301
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Reflux Esophagitis (RE)
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JP-1366 Tablets (Experimental): 20 mg qd, last for 4-8 weeks
  Interventions: Drug: Esomeprazole Magnesium (Nexium) simulation tablets
- Esomeprazole magnesium Enteric Tablets (Active Comparator): 40 mg qd, last for 4-8 weeks
  Interventions: Drug: JP-1366 simulation tablets

INTERVENTIONS:
Drug: JP-1366 simulation tablets — qd, last for 4-8 weeks
  Arms: Esomeprazole magnesium Enteric Tablets
Drug: Esomeprazole Magnesium (Nexium) simulation tablets — qd, last for 4-8 weeks
  Arms: JP-1366 Tablets

SUMMARY:
To evaluate the efficacy and safety of JP-1366 tablets and Nexium® (Esomeprazole magnesium enteric-coated tablets) in subjects with reflux esophagitis.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of JP-1366 tablets and Nexium® (Esomeprazole magnesium enteric-coated tablets) in subjects with reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign a written informed consent form, and be able to understand the information provided and comply with the program requirements;
2. Age between 18-75 years old (including boundary values) during screening, both male and female are acceptable.
3. Those who have experienced heartburn and reflux symptoms (with medical records) within 7 days before screening or who have been diagnosed with reflux esophagitis by endoscopic examination within 7 days before screening;
4. Screening period for upper gastrointestinal endoscopy, diagnosed with grade A-D reflux esophagitis in Los Angeles (those who have received endoscopic examination results from our center, have been judged by researchers to meet the diagnostic criteria, and have not been examined within 14 days before randomization, do not need to repeat this examination).
5. LA-A level subjects, esophageal reflux monitoring during the screening period, acid exposure time percentage > 4%;
6. Women of childbearing age or significant other male subjects of childbearing age are willing to use effective contraceptive measures throughout the study period, such as oral, implanted, or injected contraceptive hormones, or use mechanical products such as intrauterine devices or barrier methods (uterine caps, , spermicides), or practice abstinence or self/significant other sterilization (such as vasectomy, hysterectomy, bilateral salpinectomy, or bilateral oophorectomy).

Exclusion Criteria:

1. Known to be allergic to the test drug and any of its components or to esomeprazole magnesium and its components;
2. Those who cannot accept upper gastrointestinal endoscopy;
3. Patients with gastroesophageal varices, hiatal hernia, Zollinger-Ellison syndrome, achalasia, irritable bowel syndrome or inflammatory bowel disease;
4. History of eosinophilic esophagitis and Barrett's esophagus (≥ 3cm), confirmed by upper gastrointestinal endoscopy during the screening period;
5. Screening for patients with active peptic ulcers and active upper/lower gastrointestinal bleeding within the first 3 months; or patients with a history of active peptic ulcers and active upper/lower gastrointestinal bleeding more than 3 months after screening, and those who did not recover after endoscopic examination of the upper gastrointestinal tract during the screening period;
6. Patients with concomitant diseases that may affect esophageal motility (such as scleroderma, viral infection or fungal infection, etc.), or those with a history of esophageal radiotherapy or cryotherapy;
7. Have undergone surgery to reduce gastric acid secretion, or any surgery that affects the structure or function of the esophagus, stomach, or duodenum (except for benign tumor resection, benign polyp endoscopic resection, simple suture surgery such as gastric perforation);
8. Subjects with warning symptoms of upper gastrointestinal malignancies or gastrointestinal malignancies (such as swallowing pain, severe dysphagia, bleeding, weight loss, anemia, hemoptysis or hematochezia) (except for those with negative endoscopic malignancies);
9. People with a history of the following clinically significant diseases:

Those with a history of hemorrhagic stroke or any of the following intracranial diseases (bleeding, tumors, arteriovenous malformations (AVMs), or aneurysms); There are recurrent upper gastrointestinal or gastrointestinal ulcers/bleeding, and researchers believe that there is an increased risk of bleeding or clinical bleeding has occurred within the past 6 months before screening.

Those who have had acute clinical hepatitis or a history of major liver disease (active phase of chronic hepatitis, cirrhosis, or chronic liver dysfunction) within the past year before screening.

Screening for those who have had myocardial infarction, acute coronary syndrome, viral myocarditis, or pulmonary embolism within the past 6 months; those who have undergone coronary artery revascularization within 6 months; transient ischemic attack or ischemic stroke.

Patients with a history of chronic congestive heart failure and NYHA IV heart function.

There are severe arrhythmias that require treatment with Class Ia or III antiarrhythmic drugs; arrhythmias with diseased sinus syndrome, Class II or III atrioventricular block, and pacemakers have not yet been implanted.

People with a history of prolonged QTc interval or screening period with QTc interval ≥ 480ms (according to Fridericia correction formula, where QTc = QT/RR ^ 0.33).

Subjects with any history of active malignant tumors within the first 5 years of screening (excluding cured basal cell carcinoma, papillary thyroid carcinoma, and radical resection of carcinoma in situ such as intraductal carcinoma of the and cervical carcinoma in situ).

Subjects who need to continue receiving non-steroidal anti-inflammatory drugs (such as aspirin), systemic corticosteroids, or antithrombotic drugs during the trial period (excluding those who use prophylactic low-dose aspirin (≤ 100mg/day)).

12. Subjects who have taken gastric acid inhibitors (e.g. P-CAB, PPI) within 2 weeks before the first dose; or subjects who have taken H2 receptor blockers within 1 week before the first dose; 13. Subjects who were using retroviral antiviral drugs such as azanavir and nefinavir at the time of screening; 14. Those who meet any of the following requirements during the screening: Serum creatinine > 1.5 × ULN; history of chronic kidney disease, estimated glomerular filtration rate (eGFR) < 30ml/min/1.73m2.

Total bilirubin > 1.5 × ULN, alanine aminotransferase (AST)/aspartate aminotransferase (ALT) > 3 × ULN.

15. Have participated in any systemic therapeutic drug clinical trial (defined as administered) within the first 3 months of screening or within 5 half-lives of the test drug (whichever is longer); 16. Pregnant or lactating women; 17. The investigator determines that the subjects are not suitable to participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with esophageal mucosal healing confirmed by upper gastrointestinal endoscopy within 8 weeks of treatment | Week 4-8

SECONDARY OUTCOMES:
Percentage of subjects with esophageal mucosal healing confirmed by upper gastrointestinal endoscopy within 4 weeks of treatment | Week 0-4
Changes in the severity of major symptoms (heartburn and reflux) compared to the base line at 4 and 8 weeks after treatment. | Week 0-4 and week4-8
Changes in the frequency of major symptoms (heartburn and reflux) compared to the base line at 4 and 8 weeks after treatment. | Week 0-4 and week4-8
Changes in the overall score of gastroesophageal reflux disease health-related quality of life (GERD-HRQL) compared to the base line at 4 and 8 weeks after treatment | Week 0-4 and week4-8
  evalutated by Gastroesophageal reflux disease health-related quality of life(GERD-HRQL), the value is [-50,0] and the lower score means better outcome.
The proportion of positive answers to "treatment satisfaction" in the GERD-HRQL scale | Week 0-8
  evalutated by Gastroesophageal reflux disease health-related quality of life(GERD-HRQL), it was measured by the proportion of postive answers of overall popultation
Changes in RDQ questionnaire scores compared to the base line at 4 and 8 weeks after treatment | Week 0-4 and week4-8
  evaluated by reflux disease questionnaire(RDQ), the value is [-40,0] and the lower scorce means better outcome.
Number of participants with treatment-related adverse events of Treatment and Control groups as assessed by CTCAE v4.0 | Week0-5 or Week 0-9

OTHER OUTCOMES:
Percentage of subjects without major symptoms (heartburn and reflux) occurring within 1 week, 4 weeks, and 8 weeks after treatment (day, night, day, and night). | Week0-4 or Week0-8
Percentage of days without major symptoms (heartburn and reflux) occurring within 1 week, 4 weeks, and 8 weeks after treatment (day, night, day, and night) | Week0-4 or Week0-8
The first time there were no major symptoms (heartburn and reflux) for 7 consecutive days after treatment | Week0-4 or Week0-8

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical Universtiy, Beijing, Beijing Municipality, China